CLINICAL TRIAL: NCT02010827
Title: Endogenous Glucoseproduction in Patients With Type 2 Diabetes Mellitus During Oral Glucose and iv. Glucose Infusion
Acronym: EGP_Glucagon
Status: Completed | Type: Observational
Sponsor: University Hospital, Gentofte, Copenhagen (Other)
Responsible Party: Principal Investigator, Asger Lund, MD, University Hospital, Gentofte, Copenhagen
Other Study IDs: H-4-2013-012
Record Dates: First submitted 2013-11-27; First posted 2013-12-13 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-11

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Diabetes mellitus; Glucagon; Endogenous glucose production; Incretin hormones
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Glucose Tolerance Test

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — hole blood, serum, white cells, urine
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Patients: Patients
  Interventions: Biological: isoglycemic intravenous glucose infusion and Glucagon infusion, day C; Biological: Oral glucose tolerance test, day A; Biological: intravenous iv glucose infusion, day B
- healthy controls: healthy controls
  Interventions: Biological: isoglycemic intravenous glucose infusion and Glucagon infusion, day C; Biological: Oral glucose tolerance test, day A; Biological: intravenous iv glucose infusion, day B

INTERVENTIONS:
Biological: isoglycemic intravenous glucose infusion and Glucagon infusion, day C — Infusion of 0.8ng/kg/min glucagon from time 0-25min
Biological: Oral glucose tolerance test, day A
Biological: intravenous iv glucose infusion, day B

SUMMARY:
We want to investigate how lack of glucagon suppression during an oral glucose tolerance test in patients with type 2 diabetes contributes to patients postprandial hyperglycemia.

DETAILED DESCRIPTION:
Patients with type 2 diabetes mellitus (T2DM) are not able to suppress their glucagon secretion after a meal or after ingestion of glucose. Previous studies have shown that gastrointestinal hormones might play a role in this phenomenon. However, it has not yet been possible to determine whether this lack of glucagon suppression postprandially results in an increased endogenous glucose secretion, and thus is a factor in the patients postprandial hyperglycemia.

We aim to perform oral glucose tolerance tests and isoglycemic intravenous glucose infusions with and without a continuous glucagon infusion in patients with T2DM and healthy control subjects. The glucagon infusion is aiming at copying the inappropriate "physiological" glucagon response observed in patients with T2DM.

ELIGIBILITY:
Inclusion Criteria:

Patients with T2DM

* Caucasions above 35 years of age with diet and/or tablettreated T2DM of at -least three months (diagnosis acording to WHO)
* Normal haemoglobin
* Informed consent

Healthy Subjects

* Normal fasting plasma glucose (FPG) and normal HbA1C (according to the -World Health Organization (WHO) criteria)
* Normal haemoglobin
* Age above 35 years
* Informed consent

Exclusion Criteria:

* Inflammatory bowel disease
* Nephropathy (serum creatinine >150 µM and/or albuminuria)
* Severe liver disease (serum alanine aminotransferase (ALAT) and/or serum aspartate aminotransferase (ASAT) >3×normal values)
* Pregnancy and/or breastfeeding
* Age above 80 years
* Any condition that the investigator feels would interfere with trial participation

Patients with T2DM

Healthy Subjects

* Diabetes mellitus (DM)
* Prediabetes (impaired glucose tolerance and/or impaired FPG)
* First degree relatives with DM
* Inflammatory bowel disease
* Intestinal resection and/or ostomy
* Nephropathy (serum creatinine >150 µM and/or albuminuria
* Liver disease (ALAT and/or serum ASAT >2×normal values)
* Pregnancy and/or breastfeeding
* Age above 80 years
* Any condition that the investigator feels would interfere with trial participation

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with type 2 diabetes Healthy control subjects
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2013-11; Primary Completion 2014-09 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Differences in Endogenous glucose production during the three days measured as total Area under the curve (tAUC) | Endogenous glucose production will be calculated based on blood samples at time points: -30,-15,0,10,20,30,50,70,90,120,150,180 and 240 min on all days.
  calculated based on infusions of stable isotope marked glucose

SECONDARY OUTCOMES:
Differences in glucagon during the three days measured as total Area under the curve (tAUC) | Glucagon will be measured at time points: -30,-15,0,10,20,30,50,70,90,120,150,180 and 240 min on all days.
Differences in incretin hormone levels during the three days measured as total Area under the curve (tAUC) | incretin hormone levels will be measured at time points: -30,-15,0,10,20,30,50,70,90,120,150,180, 240 min on all days.
  GIP and GLP-1
Differences in gastrointestinal hormones during the three days measured as total Area under the curve (tAUC) | At the end of the study
differences in appetite, hunger, satiety between the three days | Satiety, hunger and appetite will be measured at time points:0,30,60,90,120,150,180, 240 min during each day.
  Will be measured with visual analogue scales (VAS)

CONTACTS AND LOCATIONS:
Locations (1):
- Diabetes Research Division, University Hospital Gentofte, Hellerup, Denmark

REFERENCES:
- [Derived] Lund A, Bagger JI, Christensen M, Grondahl M, van Hall G, Holst JJ, Vilsboll T, Knop FK. Higher Endogenous Glucose Production During OGTT vs Isoglycemic Intravenous Glucose Infusion. J Clin Endocrinol Metab. 2016 Nov;101(11):4377-4384. doi: 10.1210/jc.2016-1948. Epub 2016 Aug 17. PMID 27533305